CLINICAL TRIAL: NCT01134666
Title: An Observational Study to Evaluate the Safety and Efficacy of FOLFIRI / FOLFOX Plus Cetuximab as First-line Therapy in Patients With KRAS Wild-type Metastatic Colorectal Cancer
Status: Terminated | Type: Observational
Why Stopped: The study was discontinued due to slow recruitment and subjects not completing follow up period.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Ltd., India (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 062202-517
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal neoplasms; Intestinal neoplasms; Neoplasms; cetuximab; Erbitux
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Neoplasms; Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood and Tissue

INTERVENTIONS:
Drug: Cetuximab — FOLFOX Oxaliplatin 100 mg/ m2 day 1 Folinic Acid 400 mg/m² (racemic) or 200 mg/m² (L-form) day 1 5- FU 400 mg/m² bolus on day 1 followed by a 46-hour continuous infusion of 2,400 mg/m² day 1 FOLFIRI Irinotecan 180 mg/ m2 day 1 Folinic Acid 400 mg/m² (racemic) or 200 mg/m² (L-form) day 1 5- FU 400 mg/m² bolus on day 1 followed by a 46-hour continuous infusion of 2,400 mg/m² day 1 CETUXIMAB Cetuximab administered at loading dose of 400 mg/m2/week over 120 min followed by maintenance dose of 250 mg/m2/ week over 60 min, till disease progression or dose limiting toxicity
  Other Names: Erbitux

SUMMARY:
This is an open-label, non-randomized, prospective, multicentric, Phase IV study evaluating FOLFIRI/ FOLFOX plus cetuximab in the first-line therapy of subjects with KRAS wild-type metastatic CRC.

DETAILED DESCRIPTION:
Cetuximab, a chimeric immunoglobulin G1 (IgG1) monoclonal antibody, has been found to potentiate the effects of chemotherapy and radiotherapy in experimental systems. The findings from clinical trials suggest a favorable risk-benefit ratio of the combination of irinotecan or oxaliplatin, infusional 5-FU/FA and biweekly cetuximab, and support the current study to demonstrate the therapeutic value of the biweekly cetuximab regimen as a combination partner for those regimens in subjects with KRAS wild-type mCRC in the first-line setting. The purpose of this study is to generate post marketing surveillance (PMS) data for cetuximab in first-line mCRC, which is mandated by the Licensing Authorities.

This is an open-label, non-randomized, prospective, multicentric Phase IV study evaluating FOLFIRI/ FOLFOX plus cetuximab in the first-line therapy of subjects with KRAS wild-type metastatic CRC. The study plans to enroll 100 subjects with KRAS wild type CRC at 20 centres across India. Tumour status, physical and laboratory examinations will be performed during the baseline visit. Subjects will be administered FOLFIRI/ FOLFOX and cetuximab according to the clinical condition in the following treatment visits. Regular safety assessments and all adverse events (AEs) will be documented throughout and until the end-of-study visit. The outcome of AEs ongoing at the final tumour assessment visit will be followed up at the end-of-study visit (If possible, 6 weeks after the last administration of study medication but before second-line anticancer treatment, and not earlier than 30 days after the end of study treatment). Skin toxicity present at the end-of-study visit will be followed up until outcome is known.

OBJECTIVES

Primary Objective:

* To evaluate the safety and tolerability of Cetuximab in combination with standard chemotherapy such as FOLFOX or FOLFIRI as first-line therapy of patients with KRAS wild-type metastatic colorectal cancer.

Secondary Objective:

* To evaluate the efficacy of Cetuximab in combination with standard chemotherapy as first-line therapy of patients with KRAS wild-type metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically confirmed, adenocarcinoma of the colon or rectum (mCRC)
* Subjects with KRAS wild-type status of tumour tissue
* Chemotherapy naïve subjects
* Subject who have signed written informed consent (as per institutional protocol)

Exclusion Criteria:

* As per summary of product characteristics of cetuximab

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with KRAS wild-type CRC receiving FOLFOX/FOLFIRI and cetuximab in India.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2009-11-30 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2014-08-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability evaluated based on the incidence and severity of AEs. | From baseline to follow-up visit for any ongoing AEs

SECONDARY OUTCOMES:
Response rate | Baseline to End-of-Study Visit
  Disease Control Rate (DCR), Progression Free Survival (PFS)and Overall Survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Rana, MD, Study Director — Merck Ltd., India
Locations (40):
- India (40):
  - Indo- American Cancer Institute & Research Centre, Hyderabad, Andhra Pradesh
  - NVS Ramakrishna's Clinic, Hyderabad, Andhra Pradesh
  - Dr. Nikhil's Clinic, Secunderabad, Andhra Pradesh
  - Nikhil Gharyalpatil's Clinic, Secunderabad, Andhra Pradesh
  - Ravi Kumar's Clinic, Hyderabad, Andrapradesh
  - Ambaa Hospitals, Hyderabad, Andrapradesh
  - Swarna Sai Hospital, Hyderabad, Andrapradesh
  - Manipal Centre For Clinical Research, Mangalore, Bangalore
  - Medical College Calicut, Kerala, Calicut
  - Hemato Oncology Clinic, Ahmedabad, Gujarat
  - SKIMS, Srinagar, Jammu and Kashmir
  - S. K. I. M. S., Srinagar, Jammu and Kashmir
  - Kattimani Oncology Clinic, Hubli, Karnataka
  - Dr. T. P. Sahoo's Clinic, Bhopal, Madhya Pradesh
  - BND Onco Centre, Mumbai, Maharashtra
  - Joy Hospital, Mumbai, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Grace Nursing Home, Aizawl, Mizoram
  - Lilavati Hospital, Bandra, Mumbai
  - S.L.Raheja Hospital, Mahīm, Mumbai
  - Apollo Cancer Institute, Delhi, New Delhi
  - Rajiv Gandhi Cancer Institute & Research, Delhi, New Delhi
  - Fortis Escorts Hospital, Amritsar, Punjab
  - Dr. Rajeev Bedi's Clinic, Chandigarh, Punjab
  - D.M.C Hospital, Ludhiana, Punjab
  - IVY Hospital, Mohali, Punjab
  - Cancer Clinic, Jaipur, Rajasthan
  - SMS Hospital, Jaipur, Rajasthan
  - Bhagwan Mahaveer Cancer Hospital, Jaipur, Rajasthan
  - Bhagwan Mahaveer Cancer Hospital & Research Centre, Jaipur, Rajasthan
  - Vyas Cancer Care, Jodhpur, Rajasthan
  - TC 14/ 764 Sreemangalam, Trivandrum, Tamil Nadu
  - Shati Gopal Hospital, Ghaziabad, Uttar Pradesh
  - Annapurna Medical and Cancer Relief Society, Lucknow, Uttar Pradesh
  - Chittaranjan National Cancer Institute, Kolkata, West Bengal
  - Apollo Gleneagles Cancer Hospital, Kolkata, West Bengal
  - Nothern Railway Central Hospital, Delhi
  - Indraprastha Apollo Hospital, Delhi
  - Shanti Mukand Hospital, Delhi
  - Dharamshila Cancer Hospital & Research Centre, Delhi